CLINICAL TRIAL: NCT01050140
Title: The Metabolic Effects of a High Fructose Versus a High Glucose Diet in Overweight Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D/10/2009
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Hepatic Fatty Acid Metabolism; Systemic Insulin Resistance; Oxidative Stress; Cardiovascular Status
Keywords: fructose; fatty liver disease; diet
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fructose (Experimental): 25% dietary energy from fructose
  Interventions: Dietary Supplement: high sugar diet
- glucose (Active Comparator): 25% dietary energy from glucose
  Interventions: Dietary Supplement: high sugar diet

INTERVENTIONS:
Dietary Supplement: high sugar diet — 25% of dietary energy from fructose or glucose

SUMMARY:
Dietary consumption of fructose has increased by nearly 50% since 1960.

A high fructose diet (HFrD) results in greater visceral adiposity and systemic insulin resistance than a high glucose diet. The effects of fructose on liver fatty acid and ATP stores, systemic oxidative stress and cardiovascular status are not fully known.

DETAILED DESCRIPTION:
The protocol will assess the following outcomes:

1. The ultimate fate of this increased hepatic fatty acid production following a high fructose vs. glucose diet
2. The effect of a high fructose vs. glucose diet on liver ATP stores
3. The effect of a high fructose vs. glucose diet on markers of oxidative stress
4. The effect of a high fructose vs. glucose diet on cardiovascular status

Factors critical to carbohydrate metabolism such as systemic insulin resistance, body composition, energy expenditure, physical activity will also be assessed.

32 centrally overweight healthy males with a low baseline fructose intake will be recruited. They will be randomised double blindly to receive 25% of their dietary energy requirements from either fructose or glucose for 14 days.

The sugars will first be taken in an energy balanced and then an overfeeding setting.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index 25-32
2. Waist > hip circumference
3. Age 18-50 years
4. Male

Exclusion Criteria:

1. Reported weight change > 3 kg in prior 3/12
2. Active health problems
3. Contraindications to MRI scanning
4. Symptoms of functional bloating or irritable bowel syndrome
5. Abnormal liver or renal function tests
6. Random glucose greater than 11.0 mmol/L
7. Evidence of metabolic or viral liver disease as screened for by hepatitis B and C serology, and ferritin.
8. Alcohol intake > 21 units per week
9. Vegetarianism
10. Normal daily fructose intake from drinks greater than that in 500ml of coca cola
11. Abnormal carbohydrate energy contribution to baseline diet - defined as greater than 2 standard deviations from the mean of the National Diet and Nutrition Survey 2002 data

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Liver triglyceride content | 2 weeks

SECONDARY OUTCOMES:
Muscle triglyceride content | 2 weeks
Total abdominal visceral fat content (MRI) | 2 weeks
Liver ATP, PME concentration and pH (31P MRS) | 2 weeks
Liver de novo lipogenesis | 2 weeks
Resting energy expenditure, lipid and carbohydrate oxidation rates | 2 weeks
Hepatic and systemic insulin resistance | 2 weeks
Cardiovascular measures using finometry | 2 weeks
Systemic oxidative stress and inflammatory cytokine profile | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Study Chair — School of Biomedical Sciences, Nottingham University, UK; Richard D Johnston, MRCP, Principal Investigator — School of Biomedical Sciences, Nottingham University, UK
Locations (1):
- School of Biomedical Sciences, University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Johnston RD, Stephenson MC, Crossland H, Cordon SM, Palcidi E, Cox EF, Taylor MA, Aithal GP, Macdonald IA. No difference between high-fructose and high-glucose diets on liver triacylglycerol or biochemistry in healthy overweight men. Gastroenterology. 2013 Nov;145(5):1016-1025.e2. doi: 10.1053/j.gastro.2013.07.012. Epub 2013 Jul 19. PMID 23872500